CLINICAL TRIAL: NCT04200976
Title: Telephone Delivery of Cognitively Augmented Behavioral Activation (CABA) for Traumatic Brain Injury
Brief Title: Telephone Delivery of Cognitively Augmented Behavioral Activation (CABA)
Acronym: Tele-CABA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Megan Callahan, Principal Investigator, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PortlandVAMC
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Traumatic Brain Injury; Posttraumatic Stress Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-CABA (Experimental): Participants who engage in the Tele-CABA intervention.
  Interventions: Behavioral: Tele-CABA
- Usual Care (Placebo Comparator): Participants who do not engage in the Tele-CABA intervention during their time in the study. They will be eligible to receive Tele-CABA following completion of the 6-month questionnaires and cognitive assessment (as a courtesy).
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Tele-CABA — Tele-CABA uses Behavioral Activation (BA) to identify meaningful goals and activities while learning cognitive skills to aid in working toward those goals. Early sessions of Tele-CABA focus on learning about TBI and lifestyle skills that can improve thinking abilities and mood. Cognitive skills taught each week include internal and external skills to help manage problems with memory, attention, and regulation of thinking processes. Investigators and patients will spend a part of each session applying the cognitive skills to managing real life situations and getting patients active in the service of personal goals.
  The Tele-CABA intervention will be delivered over 10 weekly, 60-minute telephone sessions.
  Arms: Tele-CABA
Behavioral: Usual Care — Participants in the UC group will continue to receive their regular medical, psychiatric, and psychotherapeutic care.
  Arms: Usual Care

SUMMARY:
Traumatic brain injury (TBI) is highly prevalent and frequently comorbid among Veterans and Service Members. Many of these individuals sustain more than one TBI over the course of their military careers, often with little recovery time between exposures placing them at increased risk for persistent cognitive, psychological, and psychosocial difficulties that impact daily functioning and life satisfaction.

The short-term objective of this study is to examine the efficacy of the manualized, 10-week, telephone delivery of Tele-CABA for improving cognitive and adaptive functioning. The long-term objective of this study is to develop an accessible and acceptable intervention that can be broadly disseminated to address the complex rehabilitation needs of Veterans and Service Members. The overall goal of the Tele-CABA intervention is to reduce negative cognitive and psychiatric health outcomes for Veterans and Service Members with a history of TBI, promote personal resilience, and to design an intervention that is accessible and acceptable to patients struggling to recover from TBI.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Active Duty Service Members
* History of TBI (confirmed by TBI interview)
* Self-reported cognitive complaints (as indicated on the NSI)
* Able to communicate by telephone

Exclusion Criteria:

* Active suicidal intent
* History of bipolar disorder
* History of psychotic disorder
* Decisionally impaired
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Change in the Wechsler Adult Intelligence Scale-4th Edition, Digit Span subtest | Baseline; 12 weeks; and 6 months after baseline
  Measure of attention and working memory; scaled score range = 0-20 (mean = 10; SS below 2 SD below the mean considered impaired)
Change in the Neurobehavioral Symptom Inventory (NSI) | Baseline; 12 weeks; and 6 months after baseline
  Measure of postconcussion symptom severity; total score range = 0-88 (higher total score = worse symptoms)
Change in the Satisfaction with Life Scale (SWLS) | Baseline; 12 weeks; and 6 months after baseline
  Measure of life satisfaction; total score range = 0-35 (higher total score = more satisfied)

SECONDARY OUTCOMES:
Change in the PTSD Checklist-5 (PCL 5) | Baseline; after 12 weeks; and 6 months after baseline
  Measure of PTSD symptoms; total score range = 0-80 (higher total score = worse PTSD)
Change in the Memory Compensation Questionnaire (MCQ) | Baseline; after 12 weeks; and 6 months after baseline
  Measure of the use of strategies to improve memory relevant to daily living; total score range = 0-176 (lower total score = worse functioning)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Portland Health Care System, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No